CLINICAL TRIAL: NCT01531881
Title: Autofluorescence Detection of Oral Malignancies and Database and Biospecimen Collection to Identify Biomarkers of Head and Neck Tumor Progression
Status: Completed | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: I 66805
Record Dates: First submitted 2012-01-11; First posted 2012-02-13 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, oral mucosal and tongue brushings.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research may help dentists or surgeons to better detect areas in the mouth that are either prone to cancer or are early cancers. The earlier the detection on cancer in the mouth, the better the chance that treatment or prevention can be more effective.

ELIGIBILITY:
Inclusion Criteria:

Patients with a history of suspicious lesions or currant suspicious lesions:

* No history of CIS or HNSCC
* History of clinically suspicious oral/oral pharyngeal lesions.
* Over 21 years old
* Not actively under treatment for any other type of malignancy, except Non-Melanoma Skin Cancer (NMSC)
* Must be willing to sign consent, have AFL screening with biopsies and sample collection, must be willing to complete a social and health history questionnaire

Patients with biopsy proven dysplasia, CIS or HNSCC prior to treatment:

* Patients with biopsy proven dysplasia, CIS or HNSCC without a prior history of an antineoplastic treatment, including chemo/radiation and Photodynamic Therapy
* Biopsy performed at an outside institution and referred for evaluation for treatment, or biopsied here at RPCI and proceeding for further care.
* Over 21 years of age.
* Must be willing to sign consent, have AFL screening with biopsies and sample collection, must be willing to complete a social and health history questionnaire

Patients with clinically treated CIS or HNSCC amd no evidence of disease (NED):

* Patients with prior history of HNSCC, previously treated with either surgery alone or combination of therapy, including Head and Neck radiation, with or without chemotherapy and Photodynamic Therapy including at least 3 months following completion of definitive treatment.
* Over 21 years of age
* Must be willing to sign consent, have AFL screening with biopsies and sample collection, must be willing to complete a social and health history questionnaire

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dental clinic patients
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
to investigate whether the use of a fluorescent light in the mouth can detect precancers or early cancers that are not seen on normal clinical examination. | Once at time of consent (day 1)
  The first purpose of this activity is to investigate whether the use of a fluorescent light in the mouth can detect precancers or early cancers that are not seen on normal clinical examination.

SECONDARY OUTCOMES:
The second purpose is to collect other samples from the mouth in hopes to identify changes in the proteins and/or genes that will help identify how cancers start in the mouth. | Once at time of consent (day 1)
  The second purpose is to collect other samples from the mouth in hopes to identify changes in the proteins and/or genes that will help identify how cancers start in the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Schlecht, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States